CLINICAL TRIAL: NCT05942092
Title: A Retrospective Multicentric Clinical Study Comparing Radioguided Occult Lesion Localization (ROLL) and Magnetic Seed in the Intraoperative Localization of Non-palpable Breast Lesions During Breast Conservative Surgery.
Brief Title: ROLL Versus Magnetic Seed for Preoperative Localization of Non-palpable Breast Lesion: Comparison Between Techniques.
Acronym: SEED01
Status: Active, not recruiting | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Principal Investigator, Fabio Corsi, Professor, Istituti Clinici Scientifici Maugeri SpA
Other Study IDs: 2755
Record Dates: First submitted 2023-06-27; First posted 2023-07-12 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: Non-palpable breast lesion
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy, Segmental

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ROLL
  Interventions: Procedure: Breast conserving surgery
- SEED
  Interventions: Procedure: Breast conserving surgery

INTERVENTIONS:
Procedure: Breast conserving surgery — Breast conserving surgery after lesion's localization with ROLL or magnetic seed

SUMMARY:
Nowadays, Breast Conservative Surgery (BCS) is the standard of care for patients affected by early breast lesions. Screening programmes led to an increase of impalpable breast lesion detection rates. These patients are often eligible for BCS and an accurate preoperative localization technique for the detection of the lesion is required in order to guarantee a safe surgical excision.

The primary goal of BCS is to obtain a complete resection of the tumor with disease-free surgical margins. The presence of tumor on surgical margins on postoperative histological examination of the specimen increases the risk of local recurrence and it requires a surgical re-excision. For all these reasons different techniques for localization of occult breast lesions have been developed over time. Since '70s, the wire guided localization (WGL) technique has represented the gold standard technique; however, it has several limitations such as wire migration or fracture and patient's referred discomfort related to wire placement. Other techniques have been proposed such as the ROLL and magnetic seeds.

The ROLL consists of the injection of a radioactive substance into the breast lesion and the localization during surgery is allowed by using a handheld gamma probe. Limitations of this technique are represented by the need of radioactive injection the day before surgery with subsequent longer hospitalizations and the possible spread of the radioactive substance into breast tissue leading to larger resections.

The latest technological evolution is represented by magnetic seeds, small devices deployed into the lesion even up to more than 30 days before surgery and identified with a specific magnetic probe during surgery.

Currently there are several studies of comparison between the WGL and the more modern techniques. All of these data claim the effectiveness of the new "wire-free" methodics ensuring a safe surgical resection with tumor-free margins and, in some cases, a better aesthetic result.

Studies of comparison between the modern techniques are limited. There is no scientific evidence of the superiority of magnetic seeds compared to ROLL.

The aim of this retrospective study is to compare ROLL with magnetic seed to assess their efficacy in the localization of non-palpable breast lesions.

ELIGIBILITY:
Inclusion Criteria:

* Female patients between 18 and 85 years who underwent to breast conservative surgery for non-palpable occult breast lesions;
* Intraoperative localization of breast lesion with ROLL or magnetic seed;
* Preoperative diagnosis on histology or cytology of borderline lesion (B3 or C3) or malignant lesion (B4-B5 or C4-C5).

Exclusion Criteria:

* B2 or C2 at preoperative needle breast biopsy or fine needle breast aspiration.
* Breast tumor localization with clip for neoadjuvant chemotherapy.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer is gender based
Study Population: Breast cancer women with non-palpable lesions
Sampling Method: Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Free-surgical margins | 6 months
  Number of surgical procedures in which surgical margins are tumor disease-free ("no ink on tumor" for invasive cancer and margin of 2 mm for in situ-carcinoma).

SECONDARY OUTCOMES:
Excess breast resection | 6 months
  Excess breast resection calculated by the "calculated resection ratio" (CRR=total resection volume/optimal resection volume)
Surgery time | 6 months
  Surgery duration
Hospitalization's days | 6 months
  Number of hospitalization's days
Complications | 6 months
  Complications occurred after biopsy or surgery
Reintervention | 6 months
  Reintervention rates
Follow up | 5 years after enrollment
  5-years follow-up outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Istituti Clinici Scientifici Maugeri SpA, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No